CLINICAL TRIAL: NCT06809218
Title: INSPiRE-ICU 1 & 2: A Pooled Analysis of Long-Term Outcomes at 3 and 6 Months After Inhaled Isoflurane Delivered Via the Sedaconda ACD-S Compared to Intravenous Propofol for Sedation of Mechanically Ventilated Intensive Care Unit Adult Patients
Brief Title: A Pooled Analysis of Long-Term Outcomes After Inhaled Isoflurane Via the Sedaconda ACD-S Compared to Intravenous Propofol
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sedana Medical (Industry)
Collaborators: Critical Illness, Brain Dysfunction, and Survivorship Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SED003_SED004
Record Dates: First submitted 2025-01-08; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Post-Intensive Care Syndrome; Sedation
Keywords: Sedation; Inhaled Sedation; Long-term Outcomes; Cognitive Outcomes; INSPiRE-ICU; Post-Traumatic Stress Disorder; Activities and Daily Living; Quality of Life
MeSH Terms: conditions — postintensive care syndrome; Stress Disorders, Post-Traumatic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: For the Long-term follow-up part of the INSPiRE-ICU 1 & 2 studies, a separate centralized team at the Critical Illness, Brain Dysfunction and Survivorship (CIBS) center at Vanderbilt University Medical Center, is conducting the assessments and are not informed about the study treatment patients received at their respective site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inhaled isoflurane administered via Sedaconda ACD-S (Experimental): Intervention: isoflurane
  Interventions: Drug: Inhaled isoflurane administered by Sedaconda ACD-S
- Propofol administered as intravenous infusion (Active Comparator): Treatment: propofol
  Interventions: Drug: Intravenous infusion of propofol

INTERVENTIONS:
Drug: Inhaled isoflurane administered by Sedaconda ACD-S — Intervention: isoflurane
  Arms: Inhaled isoflurane administered via Sedaconda ACD-S
Drug: Intravenous infusion of propofol — Intervention: propofol
  Arms: Propofol administered as intravenous infusion

SUMMARY:
This pooled analysis will assess Cognitive, Mental Health, Functioning, and Quality of Life Assessments data from the Phase 3 registration studies INSPiRE-ICU 1 (NCT05312385) and INSPiRE-ICU 2 (NCT05327296) to explore potential differences in Long-Term Outcomes at 3 and 6 months after treatment between critically ill mechanically ventilated patients sedated with inhaled isoflurane compared to sedated with intravenous propofol.

The analyses were pre-planned and agreed prior to completion of enrollment of either study.

DETAILED DESCRIPTION:
SED003 and SED004 are two Phase 3 studies conducted in the US, with a goal to demonstrate non-inferiority of isoflurane administered via Sedaconda ACD-S to the current standard of care (SOC), IV propofol infusion, in patients requiring sedation and mechanical ventilation in the ICU.

These studies are therapeutic confirmatory (Phase 3), multicenter, randomized, controlled, open-label, assessor-blinded studies. Approximately 470 patients receiving mechanical ventilation and requiring continuous sedation at approximately 30 sites in total in the United States (US) will be randomized in a 1.5:1 ratio to inhaled isoflurane (administered via the Sedaconda ACD-S device) or propofol (administered via IV infusion) for sedation, respectively. In addition, approximately 3 to 5 run-in training patients per site will be enrolled. The treatment duration is expected to be at least 12 hours and may last up to 48 (±6) hours or to the time for extubation, whichever occurs first, with a follow up period of 6 months.

Patients eligible for the studies will either have planned surgery with anticipated need for sedation and mechanical ventilation in the ICU (ie, postoperative patients) for >12 hours or have already been admitted to the ICU and anticipate needing sedation and mechanical ventilation for >12 hours.

For further information about the studies, refer to INSPiRE-ICU 1 (NCT05312385) and INSPiRE-ICU 2 (NCT05327296).

In drug studies of critically ill patients, outcomes may be assessed at remote timepoints and not merely in the ICU. This is because the "success" of interventions is not defined merely by their impact in the hospital but also by their persistent effects. The CIBS Center at Vanderbilt University Medical Center will conduct the long-term outcome assessments for a subset of patients in the INSPiRE-ICU studies.

A comprehensive battery that combines tests from diverse and relevant domains of functioning and balances the need to be sufficiently challenging to patients as well as the need to be feasibly administered and well tolerated. Crucially, this battery can be given by telephone, which allows for it to be administered by the CIBS Center to individuals from around the country, regardless of which enrollment sites they are from.

A significant proportion of the enrolled patients in the two studies will not have any follow-up data due to expected mortality as well as loss to follow-up. Since the two studies (INSPiRE-ICU 1 & 2) are identical in design and long-term follow-up is standardized and centralized, pooling of the long-term outcomes allows for improved precision of analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are enrolled in INSPiRE-ICU1 (NCT05312385) or INSPiRE-ICU2 (NCT05327296) and survived to discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
To compare cognitive function 3 months post randomization in isoflurane- vs propofol-treated patients | 3 months post Randomization
  A patient is classified as cognitive impaired if the patient has a score 2 SD (or more) worse than population mean for one test or has a score 1.5 SD (or more) worse than population mean in two or more of the following tests: TICS, WAIS IV Digit Span, Hayling Sentence Completion Test, Controlled Oral Word Association, WMS IV - Immediate Memory (Adult/Older Adult) and WMS IV - Delayed Memory (Adult/Older Adult), at 3 months post randomization.
  The analysis will take into account age, sex, level of education, total IQCODE score at baseline, total SAPS total score at baseline, medical or surgical admission duration of mechanical ventilation before randomization, study drug and treatment duration as factors.

SECONDARY OUTCOMES:
To compare memory panorama from time in the ICU in isoflurane- vs propofol-treated patients | 3 months post Randomization
  Number of factual memories, memories of feelings, or delusional memories, as assessed by the ICU Memory Tool, collected at 3 months follow-up
To compare physical outcomes and trajectories at 3 and 6 months post randomization in isoflurane- vs propofol-treated patients | 3 and 6 months post Randomization
  Activities of daily living, as assessed by the Katz ADL, at 3 and 6 months post randomization. Score ranges between 0 and 6, where 0 is the worst outcome.
To compare depressive symptoms at 3 months post randomization in isoflurane- vs propofol-treated patients | 3 months post Randomization
  Depression, as assessed by PROMIS Depression questionnaire, at 3 months post randomization
To compare anxiety symptoms at 3 months post randomization in isoflurane- vs propofol-treated patients | 3 months post Randomization
  Anxiety symptoms, as assessed by PROMIS Anxiety questionnaire, at 3 months post randomization
To compare post-traumatic stress symptoms at 3 months post randomization in isoflurane- vs propofol-treated patients | 3 months post Randomization
  Post-traumatic stress symptoms, as assessed by IES-R, at 3 months post randomization
To compare quality of life at 3 months post randomization in isoflurane- vs propofol-treated patients | 3 months post Randomization
  Quality of life at 3 months post-randomization, as assessed by WHODAS 2.0

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sackey, MD, PhD, Study Chair — Chief Medical Officer
Locations (1):
- The Critical Illness, Brain Dysfunction and Survivorship (CIBS) Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Shehabi Y, Howe BD, Bellomo R, Arabi YM, Bailey M, Bass FE, Bin Kadiman S, McArthur CJ, Murray L, Reade MC, Seppelt IM, Takala J, Wise MP, Webb SA; ANZICS Clinical Trials Group and the SPICE III Investigators. Early Sedation with Dexmedetomidine in Critically Ill Patients. N Engl J Med. 2019 Jun 27;380(26):2506-2517. doi: 10.1056/NEJMoa1904710. Epub 2019 May 19. PMID 31112380
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Mehta S, Burry L, Cook D, Fergusson D, Steinberg M, Granton J, Herridge M, Ferguson N, Devlin J, Tanios M, Dodek P, Fowler R, Burns K, Jacka M, Olafson K, Skrobik Y, Hebert P, Sabri E, Meade M; SLEAP Investigators; Canadian Critical Care Trials Group. Daily sedation interruption in mechanically ventilated critically ill patients cared for with a sedation protocol: a randomized controlled trial. JAMA. 2012 Nov 21;308(19):1985-92. doi: 10.1001/jama.2012.13872. PMID 23180503
- [Background] Sackey PV, Martling CR, Carlsward C, Sundin O, Radell PJ. Short- and long-term follow-up of intensive care unit patients after sedation with isoflurane and midazolam--a pilot study. Crit Care Med. 2008 Mar;36(3):801-6. doi: 10.1097/CCM.0B013E3181652FEE. PMID 18431266
- [Background] Mesnil M, Capdevila X, Bringuier S, Trine PO, Falquet Y, Charbit J, Roustan JP, Chanques G, Jaber S. Long-term sedation in intensive care unit: a randomized comparison between inhaled sevoflurane and intravenous propofol or midazolam. Intensive Care Med. 2011 Jun;37(6):933-41. doi: 10.1007/s00134-011-2187-3. Epub 2011 Mar 29. PMID 21445642
- [Background] Meiser A, Volk T, Wallenborn J, Guenther U, Becher T, Bracht H, Schwarzkopf K, Knafelj R, Faltlhauser A, Thal SC, Soukup J, Kellner P, Druner M, Vogelsang H, Bellgardt M, Sackey P; Sedaconda study group. Inhaled isoflurane via the anaesthetic conserving device versus propofol for sedation of invasively ventilated patients in intensive care units in Germany and Slovenia: an open-label, phase 3, randomised controlled, non-inferiority trial. Lancet Respir Med. 2021 Nov;9(11):1231-1240. doi: 10.1016/S2213-2600(21)00323-4. Epub 2021 Aug 26. PMID 34454654
- [Background] Kong KL, Willatts SM, Prys-Roberts C. Isoflurane compared with midazolam for sedation in the intensive care unit. BMJ. 1989 May 13;298(6683):1277-80. doi: 10.1136/bmj.298.6683.1277. PMID 2500195
- [Background] Chanques G, Constantin JM, Devlin JW, Ely EW, Fraser GL, Gelinas C, Girard TD, Guerin C, Jabaudon M, Jaber S, Mehta S, Langer T, Murray MJ, Pandharipande P, Patel B, Payen JF, Puntillo K, Rochwerg B, Shehabi Y, Strom T, Olsen HT, Kress JP. Analgesia and sedation in patients with ARDS. Intensive Care Med. 2020 Dec;46(12):2342-2356. doi: 10.1007/s00134-020-06307-9. Epub 2020 Nov 10. PMID 33170331
- [Background] Jerath A, Ferguson ND, Cuthbertson B. Inhalational volatile-based sedation for COVID-19 pneumonia and ARDS. Intensive Care Med. 2020 Aug;46(8):1563-1566. doi: 10.1007/s00134-020-06154-8. Epub 2020 Jun 25. PMID 32588067
- [Background] Bellgardt M, Bomberg H, Herzog-Niescery J, Dasch B, Vogelsang H, Weber TP, Steinfort C, Uhl W, Wagenpfeil S, Volk T, Meiser A. Survival after long-term isoflurane sedation as opposed to intravenous sedation in critically ill surgical patients: Retrospective analysis. Eur J Anaesthesiol. 2016 Jan;33(1):6-13. doi: 10.1097/EJA.0000000000000252. PMID 25793760
- [Background] Hughes CG, Mailloux PT, Devlin JW, Swan JT, Sanders RD, Anzueto A, Jackson JC, Hoskins AS, Pun BT, Orun OM, Raman R, Stollings JL, Kiehl AL, Duprey MS, Bui LN, O'Neal HR Jr, Snyder A, Gropper MA, Guntupalli KK, Stashenko GJ, Patel MB, Brummel NE, Girard TD, Dittus RS, Bernard GR, Ely EW, Pandharipande PP; MENDS2 Study Investigators. Dexmedetomidine or Propofol for Sedation in Mechanically Ventilated Adults with Sepsis. N Engl J Med. 2021 Apr 15;384(15):1424-1436. doi: 10.1056/NEJMoa2024922. Epub 2021 Feb 2. PMID 33528922
- [Background] Krannich A, Leithner C, Engels M, Nee J, Petzinka V, Schroder T, Jorres A, Kruse J, Storm C. Isoflurane Sedation on the ICU in Cardiac Arrest Patients Treated With Targeted Temperature Management: An Observational Propensity-Matched Study. Crit Care Med. 2017 Apr;45(4):e384-e390. doi: 10.1097/CCM.0000000000002185. PMID 27941501
- [Background] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- See also: Isoflurane 100% inhalation vapour, liquid. Summary of product characteristics. West Drayton, United Kingdon. Piramal Critical Care Ltd. Electronic medicines compendium(emc), last updated 29 October 2019. Accessed 09 September 2020. — http://www.medicines.org.uk/emc/product/9800/smpc#gref